CLINICAL TRIAL: NCT05448391
Title: An Open-label, Single-arm, Phase 2 Study to Evaluate the Safety and Efficacy of RIST4721 in Subjects With Familial Mediterranean Fever
Brief Title: A Study to Evaluate RIST4721 in Familial Mediterranean Fever (FMF)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to safety findings in other ongoing Phase 2 trials.
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIST4721-212
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- RIST4721 400 mg (Experimental): RIST4721 400 mg: 4 active (100 mg) tablets once daily for 12 weeks
  Interventions: Drug: RIST4721

INTERVENTIONS:
Drug: RIST4721 — RIST4721 tablets, 100 mg are blue, oval, biconvex film-coated tablets

SUMMARY:
A 12-week Open-label, Single-arm, Phase 2 Study to Evaluate the Safety and Efficacy of RIST4721 in Subjects with Familial Mediterranean Fever followed by an additional Open-label Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 FMF disease but no active flare at the time of screening according to Tel Hashomer criteria or EUROFEVER/Paediatric Rheumatology International Trials Organization (PRINTO) criteria for FMF
* Documented to be heterozygous or homozygous for at least one of the known clearly pathogenic MEFV gene exon 10 mutations
* Males and females must be willing to use birth control as indicated

Exclusion Criteria:

* Breastfeeding or pregnant
* Known immunodeficiency or subject is immunocompromised
* Active/latent infection with HBV, HCV, HIV, SARS-CoV-2 or TB

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious TEAEs | Baseline to Week 12

SECONDARY OUTCOMES:
Proportion of responders who achieve resolution of their index flare after initiating study treatment and do not experience a new flare from the time of resolution of the index flare until Week 12 | Baseline to Week 12

IPD SHARING:
Plan to Share IPD: No